CLINICAL TRIAL: NCT06432829
Title: Study on the Efficacy and Differential Usability of the Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders in Spanish University Students
Brief Title: Study on the Effectiveness and Differential Usability of the UP in Spanish University Students
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Sanitaria Aragón (Other)
Responsible Party: Principal Investigator, Jorge Javier Osma López, Principal Investigator, Instituto de Investigación Sanitaria Aragón
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IPES/PU-E/2024
Record Dates: First submitted 2024-05-22; First posted 2024-05-29 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Emotional Disorder; Depression, Anxiety; Emotion Regulation
Keywords: Emotional Disorders; University Students; Unified Protocol; Blended format; Online interventions; Group formats
MeSH Terms: conditions — Depression; Anxiety Disorders; Emotional Regulation

STUDY DESIGN:
Intervention Model Description: Participants will be recruited through the Psychological Care Unit (UNAP) of the University of Cordoba (Spain). The UNAP will refer to the research team those persons whose reason for consultation refers to an emotional problem (anxious and/or depressive symptomatology). Potential participants will be contacted by the research team via email and will be sent an information sheet about the study and informed consent, which they will be able to read and sign online through a Google Forms link.
Who Masked: Participant
Masking Description: Participants are informed of the assigned intervention condition before the start of the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UP in online group format (Active Comparator): The participants assigned to this condition will receive the UP in group format through 8 sessions of 2 hours duration, once a week, in online format through the Google Meet platform. Participants will receive a brief manual with the important contents of each session, the exercises to be performed and the corresponding records.
  Interventions: Behavioral: Unified Protocol for the transdiagnostic treatment of emotional disorders
- UP in blended format (UP online group + UP App) (Experimental): Participants assigned to this condition will receive the PU in a blended group format (4 online group sessions, of two hours duration in modules 1,4,6 and 7 of the PU + autonomous work through the UP-APP). Thus, participants will receive a combined intervention format, working some contents in online group sessions and others through the PU-APP.
  Interventions: Behavioral: Unified Protocol for the transdiagnostic treatment of emotional disorders

INTERVENTIONS:
Behavioral: Unified Protocol for the transdiagnostic treatment of emotional disorders — This intervention focuses on a wide range of emotional psychopathology, allowing care for comorbid disorders and subclinical or unspecified symptoms, which reduces treatment times and costs, and improves response to treatment. The intervention will be carried out in an online-group format. For ethical reasons, if any of the patients feel uncomfortable during the study with the online-group format, will may leave the group and receive individual attention. The study plans follow-ups at 1 and 3 months after the end of the treatment.

SUMMARY:
The present study seeks to compare and analyze the degree of usefulness, acceptability and implementation of the Unified Protocol (UP) in its application in two cost-effective formats, the online group and the blended online group for the treatment of emotional disorders in university students in Spain.

DETAILED DESCRIPTION:
Introduction: Emotional Disorders (EDs) are the most common disorders among the young population. Despite their high prevalence in university students, data suggest that only 16.4% of students suffering from a mental health disorder receive treatment. Therefore, the present study seeks to compare and analyze the degree of usefulness, acceptability and implementation of the Unified Protocol (UP) in its application in two cost-effective formats, the online group and the Blended online group.

Method: The study population will be university students who meet diagnostic criteria for EDs. We estimate a sample of 70 students, 35 per condition. The intervention will consist of the application of the 8 modules of the UP in two formats: online group format of 8 weekly sessions of 2 hours duration and Blended format (4 online group sessions, of two hours duration in modules 1,4,6 and 7 of the UP + autonomous work through the UP-APP). The variables evaluated will be collected before the intervention, in the post-treatment and in the follow-ups at one month and 3 months.

This study responds to the need to implement services that improve the availability and access to the treatment of EDs in the university context in Spain, and in this particular case, through the formats offered by a transdiagnostic intervention such as the UP.

ELIGIBILITY:
Inclusion Criteria:

* Be enrolled at the University of Cordoba (Spain), in any of the degrees
* Have a diagnosis of anxiety or mood disorder from the Structured Interview for Anxiety and Related Disorders, according to the DSM-5 (ADIS-5)*
* Be at least 18 years old
* Be fluent in the Spanish language
* Have a technological device (Computer, Tablet, cell phone) with internet connection
* Have a smartphone device with Android operating system
* In the case of taking pharmacological treatment for the treatment of their ED, maintenance of the same doses and medications for at least 3 months before starting their participation in the study and throughout the treatment
* Signature of the informed consent

Exclusion Criteria:

* Have a diagnosis of Obsessive Compulsive Disorder or Post Traumatic Stress Disorder
* Have a severe condition that requires priority for treatment will not be able to participate in the study. This includes a serious mental disorder (personality disorder, schizophrenia, or an organic mental disorder), suicide risk at the time of assessment, or substance abuse within the past three months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-06-15 (Estimated); Primary Completion 2024-09-15 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Structured interview for anxiety disorders and related disorders, according to the DSM-5 (ADIS-5; Brown & Barlow, 2014) | Only before of the treatment to check inclusion criteria
  Diagnostic interview to determine if the participant has a clinical diagnosis of emotional disorder (ET) and can be part of the study. The following diagnoses according to the DSM-V are included within the category of emotional disorder: major depressive disorder, dysthymic disorder, panic disorder, agoraphobia, obsessive-compulsive disorder, generalized anxiety disorder, post-traumatic stress disorder, social anxiety disorder, hypochondria, and adjustment disorders. Patients with anxiety disorders not otherwise specified and those with depressive disorders not otherwise specified will also be included in the study.
Questionnaire on Sociodemographic Data (ad hoc) | Pre-treatment data
  Information will be collected on sex, age, marital status, employment status, type of study (bachelor's degree; postgraduate: master's degree, continuing education courses; doctorate), degree taken and course in which you are enrolled.
General Depression Severity and Interference Scale (ODSIS; Bentley et al., 2014. Validated in Spanish by Osma et al., 2019) | Up to 3 months follow-up
  Evaluation through 5 items of the frequency, intensity, severity and interference of depressive symptomatology
General Severity and Interference Scale for Anxiety (OASIS; Norman et al., 2006. Validated in Spanish by Osma et al., 2019) | Up to 3 months follow-up
  Evaluation through 5 items of the frequency, intensity, severity and interference of anxious symptomatology
Multidimensional Inventory for Emotional Disorders (MEDI; Rosellini and Brown, 2019. Validated in Spanish by Osma et al., 2023) | Up to 3 months follow-up
  Evaluation through 49 items of the transdiagnostic profile of Emotional Disorders, which is composed of nine dimensions: neurotic temperament, positive temperament, depressed mood, somatic anxiety, arousal activation, social anxiety, intrusive cognitions, traumatic re-experiencing, and avoidance

SECONDARY OUTCOMES:
Emotional Regulation Difficulties Scale (DERS; Gratz and Roemer, 2004. Validated in Spanish by Hervás & Jódar, 2008) | Up to 3 months follow-up
  Evaluation through 28 items of difficulties in emotional regulation by means of 5 subscales: lack of control, rejection, interference, inattention and emotional confusion.
Emotional Regulation Questionnaire (ERQ; Gross & John, 2003. Validated in Spanish by Pineda et al., 2018) | Up to 3 months follow-up
  Evaluation of emotional regulation through 10 items, scored on a scale from 1 (strongly disagree) to 7 (strongly agree), with two subscales: cognitive restructuring and emotional suppression.
Short Version of the Five Facets of Mindfulness Questionnaire (FFMQ-SF; Bohlmeijer et al., 2011. Validated in Spanish by Asensio-Martínez et al., 2019) | Up to 3 months follow-up
  Evaluation of the five facets of mindfulness: observing, describing, acting consciously, not judging, internal experience and non-reactivity to internal experience, through 24 items.
EuroQol (Brooks, 1996. Validated in Spanish by Badia et al., 1999) | Up to 3 months follow-up
  Assessment of self-perceived health status.
Short-format Therapeutic Alliance Inventory (WAI-S; Hatcher and Gillas, 2006. Validated in Spanish by Corbella et al., 2011) | Up to 3 months follow-up
  Evaluation of the therapeutic alliance through 12 items.
Maladjustment Scale (EI; Echeburua; 2000; Validated in Spanish by Quiléz-Orden et al., in press) | Up to 3 months follow-up
  Evaluation through 6 items about the extent to which patients' psychological problems affect different areas of daily life: work or studies, social life, free time, couple relationship and family life.
An adaptation of Client Satisfaction Questionnaire (CSQ-8) of Larsen et al., 1979 | Up to 3 months follow-up
  Our adaptation includes 6 of the 8 items of the CSQ-8 (perceived quality, adequacy to previous expectations, recommendation of the treatment to friends or family, usefulness of the techniques learned, general satisfaction with the intervention and probability that they will choose an intervention of this type again) and one more item related to the discomfort generated by the intervention. Likewise, a change has been made in the Likert response scale from 4 points in the original (0 = "Bad / Not at all" to 4 = "Excellent/Very Much") to 11 in the current one (0 = "Bad / Not at all to 10 = "Excellent/Very Much").
Evaluation questionnaire of the PU modules (Ad hoc) | Up to 3 months follow-up
  Questionnaire prepared ad hoc composed of 7 questions; one of a general nature that evaluates the usefulness of the program to improve emotional regulation and six specific ones that separately evaluate the usefulness to better regulate emotions of each of the techniques that are worked on in the different modules of the PU. The response scale is Likert-type and ranges from 0 (not at all) to 10 (very much).
System Usability Scale (SUS; Brooke, 1996. Validated in Spanish by Sevilla-Gonzalez et al., 2020) | Up to 3 months follow-up
  Scale used to evaluate the usability of the app included in PU condition in hybrid online group format

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto de investigación sanitaria de Aragón, universidad de Zaragoza, Teruel, Spain

IPD SHARING:
Plan to Share IPD: Yes
Under request
Supporting Information: Study Protocol

REFERENCES:
- See also: IPES web (Investigation group) — https://ipes-group.com/